CLINICAL TRIAL: NCT04835805
Title: A Phase Ib, Open-Label, Multicenter Study to Evaluate the Safety, Pharmacokinetics, and Activity of Belvarafenib as a Single Agent and in Combination With Either Cobimetinib or Cobimetinib Plus Nivolumab in Patients With NRAS-Mutant Advanced Melanoma Who Have Received Anti-PD-1/PD-L1 Therapy
Brief Title: A Study to Evaluate the Safety and Activity of Belvarafenib as a Single Agent and in Combination With Either Cobimetinib or Cobimetinib Plus Nivolumab in Patients With NRAS-mutant Advanced Melanoma.
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO42273; 2020-003674-41 (EudraCT Number)
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — cobimetinib; Nivolumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Belvarafenib Monotherapy (Experimental): Twice daily (BID), continuous dosing.
  Interventions: Drug: Belvarafenib
- Belvarafenib Plus Cobimetinib (Experimental): Recommended dose (RD) and schedule of belvarafenib and cobimetinib selected based on the safety data, tolerability, pharmacokinetics, and anti-tumor activity tested in dose-finding phase followed by an expansion phase.
  Interventions: Drug: Cobimetinib
- Belvarafenib Plus Cobimetinib Plus Nivolumab (Experimental): Recommended dose (RD) and schedule of belvarafenib and cobimetinib plus nivolumab IV infusion every 4 weeks (Q4W) in a run-in phase followed by an expansion phase
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Belvarafenib — Twice daily (BID), continuous dosing
  Arms: Belvarafenib Monotherapy
Drug: Cobimetinib — Once daily (QD) or three times weekly (TIW) for 21 days, 7 days off
  Arms: Belvarafenib Plus Cobimetinib
Drug: Nivolumab — Once every 4 weeks (Q4W)
  Arms: Belvarafenib Plus Cobimetinib Plus Nivolumab

SUMMARY:
This study will evaluate the safety, pharmacokinetics, and activity of belvarafenib as a single agent and in combination with either cobimetinib or cobimetinib plus nivolumab in patients with NRAS-mutant advanced melanoma who have received anti-PD-1/PD-L1 therapy.

DETAILED DESCRIPTION:
The study will evaluate three treatment regimens in three arms: a belvarafenib monotherapy arm (Belva arm); a belvarafenib plus cobimetinib arm (Belva + Cobi arm) in an initial dose-finding phase followed by an expansion phase and a belvarafenib plus cobimetinib plus nivolumab arm (Belva + Cobi + Nivo arm) in a run-in phase followed by an expansion phase.

ELIGIBILITY:
Inclusion Criteria:

* ECOG Performance Status of 0 or 1
* Histologically confirmed, metastatic (recurrent or de novo Stage IV) or unresectable locally advanced (Stage III) cutaneous melanoma, that has progressed on or after treatment with anti-PD-1 or anti-PD-L1 therapy. Patients may have received up to two lines of systemic cancer therapy. Treatment with anti-PD-1/PD-L1 in the adjuvant setting is acceptable. Patients must have progressed disease at study entry
* Documentation of NRAS mutation-positive within 5 years prior to screening
* Tumor specimen availability
* Adequate hematologic and end-organ function
* Measurable disease per RECIST v1.1

Exclusion Criteria:

* Prior treatment with a pan-RAF inhibitor
* Treatment with systemic immunotherapy agents (e.g., anti-CTLA4, anti-PD(L)1, cytokine therapy, investigational therapy, etc.) within 28 days prior to C1D1
* Symptomatic, untreated, or actively progressing CNS metastases
* History or signs/symptoms of clinically significant cardiovascular disease
* Known clinically significant liver disease
* History of autoimmune disease or immune deficiency
* Prior treatment with a MEK inhibitor (cobimetinib arm)
* History of or evidence of retinal pathology on ophthalmologic examination (cobimetinib arm)
* History of immune-related AE attributed to prior anti-PD(L)1 therapy that resulted in permanent discontinuation of anti-PD(L)1 therapy (nivolumab arm)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2021-05-13 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Dose Limiting Toxicity (DLTs) | 28 Days from Cycle 1, Day 1
Percentage of Participants With Adverse Events | From Cycle 1, Day 1 Up to 4 Years
  Severity determined according to National Cancer Institute Common Terminology Criteria for Adverse Events v5.0

SECONDARY OUTCOMES:
Objective response rate (ORR) according to RECIST v1.1 | Up to Approximately 4 Years
  Defined as the percentage of participants with a CR or PR on two consecutive occasions >/= 4 weeks apart, as determined by the investigator according to RECIST v1.1
Progression free survival (PFS) according to RECIST v1.1 | Up to Approximately 4 Years
  Defined as the time from the first study treatment to the first occurrence of disease progression or death from any cause (whichever occurs first), as determined by the investigator according to RECIST v1.1
Duration of response (DOR) according to RECIST v1.1 | Up to Approximately 4 Years
  Defined as the time from the first occurrence of a confirmed objective response to disease progression or death from any cause (whichever occurs first), as determined by the investigator according to RECIST v1.1
Overall survival (OS) | Up to Approximately 4 Years
  Defined as the time from the first study treatment to death from any cause
Plasma concentration of belvarafenib at specified timepoints | Up to 30 Days After the Final Dose of Study Drug
Plasma concentration of cobimetinib at specified timepoints | Up to 30 Days After the Final Dose of Study Drug

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (17):
- United States (6):
  - California Pacific Medical Center Research Institute, San Francisco, California
  - UCSF Helen Diller Family CCC, San Francisco, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan Kettering, New York, New York
- Australia (3):
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Peter MacCallum Cancer Centre-East Melbourne, Melbourne, Victoria
  - Linear Clinical Research Ltd, Nedlands, Western Australia
- Canada (2):
  - Ottawa Hospital Regional Cancer Centre, Ottawa, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
- Germany (5):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Klinikum Mannheim GmbH Universitätsklinikum, Mannheim
  - Universitatsklinikum Tubingen, Tübingen
  - Universitätsklinikum Würzburg, Würzburg
- Asan Medical Center - PPDS, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Moschos SJ. War against NRAS-Mutant Melanoma Using Targeted Therapies Remains Challenging. Clin Cancer Res. 2022 Jul 15;28(14):2977-2979. doi: 10.1158/1078-0432.CCR-22-1256. PMID 35587446